CLINICAL TRIAL: NCT06545006
Title: Effectiveness of a Quick Release Dynamic Muscle-strengthening Program on Dynamic Stabilization of the Cervical Spine
Acronym: CERVITRAIN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL24_0006
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Rugby; Craniocerebral Trauma; Cervical Spine Injury; Stabilization
Keywords: Cervical Muscle; Dynamic Strengthening; Stabilization; Cervical Spine; Head Impact; Rugby
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Isometric Contraction

STUDY DESIGN:
Intervention Model Description: Single-center, controlled, randomized, stratified on time to activation of cervical spine extensor muscles, open-label study with blinded evaluation.
Who Masked: Investigator
Masking Description: Main Investigator will be be blinded from the group intervention. The Main Investigator will record the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Quick Release Strengthening (Experimental): The rugby player participants will do 10 sessions of 40 minutes of muscle strengthening at a rate of 2 to 3 sessions per week. 20 minutes of isometric strengthening and 20 minutes of Quick release strengthening
  Interventions: Other: isometric contractions; Other: Quick Release
- Stroboscopic Glasses Tasks (Sham Comparator): The rugby player participants will do 10 sessions of 40 minutes of muscle strengthening at a rate of 2 to 3 sessions per week. 20 minutes of exercises with a rugby ball while wearing stroboscopic glasses.
  Interventions: Other: isometric contractions; Other: stroboscopic glasses

INTERVENTIONS:
Other: isometric contractions — Participants will perform 20 minutes of isometric contractions in different positions, with contraction durations of 10 seconds and a number of repetitions between 4 and 10, depending on their progress in the training program.
Other: stroboscopic glasses — This training involves performing skill exercises with a rugby ball while wearing stroboscopic glasses. The glasses have alternating opaque and clear sections, causing multiple and/or fragmented vision.
  The goal is to improve the processing of visual information at the level of higher functions. This aids in decision-making. It does not involve the same structures and functions implicated in reflexive muscle recruitment strategies as the Quick Release, so it should not be a confounding factor. However, it provides a beneficial, stimulating, and enjoyable training session, increasing subject adherence as they work on a skill useful in their sport.
  Arms: Stroboscopic Glasses Tasks
Other: Quick Release — The distance (in mm) of the anterior head translation will be measured using a linear displacement sensor. The subject will be instructed to recruit their extensor muscles as quickly and as strongly as possible to minimise the head displacement distance. They will be aware of their score after each repetition (real-time feedback).
  Subjects must react to a rapid forward displacement of the cervical spine, without impact. To generate this forward displacement without impact, subjects are positioned with support in front of the forehead, holding their head and neck. The subject must exert an isometric flexion effort against this frontal support (energy storage), with the intensity set by the examiner based on the Maximum Isometric Force measured during a prior maximal isometric test. The frontal resistance will suddenly release, and the head displacement in the sagittal plane will be measured until the recruitment of the cervical spine extensor muscles stops this displacement
  Arms: Quick Release Strengthening

SUMMARY:
The goal of this clinical trial is to learn if Quick Release dynamic strengthening of the cervical spine extensor muscles' reflex could improve dynamic stabilisation capacities of the cervical spine by reducing muscle activation delay in amateurs rugby players. The main questions it aims to answer are described as follows:

The primary outcome measure is the comparison between the intervention and control groups of the variation in activation delay of the cervical spine extensor muscles in milliseconds (ms) between the beginning and the end of the strengthening program. The activation delay in milliseconds corresponds to the time between the onset of impact application on the head and the onset of reactive muscle force production measured by the Cervistab© ergometer.

The secondary outcomes are also a comparison between the two groups of the variations from the beginning to the end of the strengthening program for the followings parameters, measured during with the Cervistab© machine:

* Reflex Force Production Rate (N/ms): slope of the force/time graph.
* Maximum Reactive Force (N): maximum force value produced within 300 ms following impact.
* In both intervention groups: measurement of the variation in head displacement (in mm) during quick release strengthening protocol.
* In each subgroup, 10 participants will be equipped with Instrumented Mouthguards. Researchers will compare the variation in workload measured by these mouthguards during Cervistab evaluations conducted before and after the training protocol.

Researchers will compare the intervention group to a distractor (control) arm to see if our training protocol has an impact on the activation delay.

DETAILED DESCRIPTION:
Rugby authorities are seeking preventive measures to reduce cranio-cervical injuries. Literature suggests that early and strong contraction of cervical spine muscles could decrease this risk. The Quick Release principle, using maximal isometric contractions and non-impact disturbances, might improve the dynamic stabilization of the cervical spine. No study has yet evaluated the effect of muscle strengthening programs on this stabilization.

It is hypothesized that specific training of the cervical spine extensor muscles could reduce activation delay and increase reflexive force.

This study is a single-centre, controlled, randomised, and stratified based on activation delay.

It is an open study with blind evaluation. Randomization will be stratified based on the activation delay of the cervical spine extensor muscles into two sub-groups (slow and fast), measured during the Cervistab© test at the inclusion visit.

Researchers propose an open-label study with blind evaluation: The principal investigator, who will conduct the pre- and post-training protocol tests, will not be involved in the training protocol (conducted by the associated investigator) and will therefore not know which program the tested subject completed.

Both groups will undergo a foundational cervical muscle strengthening regimen, which includes classic isometric contraction strengthening (duration = 20 minutes) at the beginning of their training session.

The second part of each training session will depend on the group to which they have been randomised (also 20 minutes):

* Either 20 minutes of dynamic strengthening through Quick Release (tested arm)
* Or 20 minutes of decision-making aid with Stroboscopic Glasses (control arm with distractor)

Both groups will do 10 trainings of 40 minutes dispatched on one month.

Cervistab ergometer is a machine developped by the main investigator and engineers that records force (in newton) as a function of time. It delivers impacts over the head of the subject. Each subject puts himself in "scrum" position and take small impacts over the head and we can measure the reflex force production rate after the activation delay.

Distractor arm : The comparison group will have to do useful tasks for their rugby practice that does not have an impact on the primary outcome. Here, researchers will ask the comparison group to use stroboscopic glasses to train their decision skills in catching and throwing rugby balls. The stroboscopic glasses switch from bright to dark at a certain frequency and hence, reduce the amount of visual information.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Possess a valid rugby practice licence

Non Inclusion Criteria :

* History of serious cervical trauma during his career with : Need for surgery (in case of arthrodesis at 2 or more levels) and/or Persistent after-effects (sensory or motor), any cervicobrachial symptomatology.
* History of epileptic disease
* Any concussion less than one month old
* Population with special legal protection: Pregnant or breast-feeding woman (L. 1121-5), subject deprived of liberty (art.L. 1121-6), minors L. 1121-7, patient unable to give consent (1121-8), protected adults L. 1121-8, not affiliated to a social security scheme (L1121-8-1), vulnerable persons (L.1122-2), exclusion period (Article L1121-12).
* Refusal of consent after information
* Participant not fluent in French and without a support person able to read.
* People who practice other contact sports.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of the activation delay | Baseline and at end (week 6)
  the time between the onset of impact application on the head and the onset of reactive muscle force production (in miliseconds)
  comparison between the intervention and control groups of the variation in muscle activation delay of the cervical spine extensors (in ms) between the start and the end of the strengthening program. The activation delay in ms corresponds to the time between the start of the application of impact to the head and the start of production of reactive muscle force during the test on the Cervistab© ergometer.

SECONDARY OUTCOMES:
Rate of Reflex Force Production | Baseline and at end (week 6)
  Comparison between the 2 groups of the variations between the beginning and the end of the reinforcement program, of the following parameter : slope of the force/time graph in newton per miliseconds
Maximum Reactive Force | Baseline and at end (week 6)
  Comparison between the 2 groups of the variations between the beginning and the end of the reinforcement program, of the following parameter : maximum force value produced within 300 ms following impact in newton
Workload | Baseline and at end (week 6)
  In each subgroup of 10 participants equipped with Instrumented Mouthguards, we will compare the variation in Workload measured by these mouthguards during Cervistab evaluations conducted before and after the training protocol.(in G)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Julia, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- EuroMov Université de Montpellier, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Undecided
Researchers will make available any informations useful for reviewers or other researchers interested by doing complementary studies based on our works

REFERENCES:
- [Result] Bohu Y, Julia M, Bagate C, Peyrin JC, Colonna JP, Thoreux P, Pascal-Moussellard H. Declining incidence of catastrophic cervical spine injuries in French rugby: 1996-2006. Am J Sports Med. 2009 Feb;37(2):319-23. doi: 10.1177/0363546508325926. PMID 19182111
- [Result] Eckner JT, Oh YK, Joshi MS, Richardson JK, Ashton-Miller JA. Effect of neck muscle strength and anticipatory cervical muscle activation on the kinematic response of the head to impulsive loads. Am J Sports Med. 2014 Mar;42(3):566-76. doi: 10.1177/0363546513517869. Epub 2014 Jan 31. PMID 24488820
- [Result] Pedersen MT, Essendrop M, Skotte JH, Jorgensen K, Fallentin N. Training can modify back muscle response to sudden trunk loading. Eur Spine J. 2004 Oct;13(6):548-52. doi: 10.1007/s00586-004-0679-3. Epub 2004 Feb 25. PMID 14986074
- [Result] Garrett JM, Mastrorocco M, Peek K, van den Hoek DJ, McGuckian TB. The Relationship Between Neck Strength and Sports-Related Concussion in Team Sports: A Systematic Review With Meta-analysis. J Orthop Sports Phys Ther. 2023 Oct;53(10):585-593. doi: 10.2519/jospt.2023.11727. PMID 37428807
- [Result] Tognella F, Mainar A, Vanhoutte C, Goubel F. A mechanical device for studying mechanical properties of human muscles in vivo. J Biomech. 1997 Oct;30(10):1077-80. doi: 10.1016/s0021-9290(97)00067-5. PMID 9391877
- [Result] Daneshvar DH, Goldstein LE, Kiernan PT, Stein TD, McKee AC. Post-traumatic neurodegeneration and chronic traumatic encephalopathy. Mol Cell Neurosci. 2015 May;66(Pt B):81-90. doi: 10.1016/j.mcn.2015.03.007. Epub 2015 Mar 7. PMID 25758552